CLINICAL TRIAL: NCT03463070
Title: The Effect of Misoprostol Given Preoperative Versus Postoperative on Blood Loss With Elective Cesarean Section: Randomized Controlled Trial
Brief Title: Misoprostol Before and After Cesarean Section
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: sarah mohamed hassan (Other)
Responsible Party: Sponsor-Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1122345
Record Dates: First submitted 2018-03-04; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Post Partum Hemorrhage
Keywords: misoprostol; postpartum haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative misoprostol group (Active Comparator): 70 women who received 600 mg misoprostol rectally preoperatively before cesarean section
  Interventions: Drug: rectal misoprostol 600mg
- postoperative misoprostol group (Active Comparator): 70 women who received 600 mg misoprostol postoperatively at operating theatre after cesarean section
  Interventions: Drug: rectal misoprostol 600mg

INTERVENTIONS:
Drug: rectal misoprostol 600mg — 70 women who received 600 mg misoprostol postoperatively at operating theatre

SUMMARY:
comparison of the effect of misoprostol before and after cesarean on the blood loss

DETAILED DESCRIPTION:
70 women who received 600 mg misoprostol rectally preoperatively versus 70 women who received 600 mg misoprostol postoperatively at operating theatre

ELIGIBILITY:
Inclusion Criteria:

* Women not in active labor have reactive non-stress test.
* No contraindications to prostaglandins.
* Have no history of coagulopathy.

Exclusion Criteria:

* Placenta previa.
* Maternal hypertension.
* Diabetes mellitus.
* Previous CS and those with active labor.
* Multiple Fibroid uterus.
* Multiple pregnancies or polyhydramnios.
* Previous myomectomy, previous history of PPH.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | the operation time
  Difference in weight of linen towels (gm)+Volume of contents of suction bottle (ml)
postoperative blood loss | every 6 hours during first 24 hours.
  weighing the soaked napkins after collection of soaked towel

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No